CLINICAL TRIAL: NCT03053973
Title: Nocturnal Non-Invasive Ventilation in COPD Patients With Stable Hypercapnic Respiratory Failure: Why and in Which Patient Might This be Effective?
Brief Title: The Effects of Nocturnal Non-invasive Ventilation in Stable COPD
Acronym: RECAPTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Wijkstra (Other)
Responsible Party: Sponsor-Investigator, Peter Wijkstra, Prof. Dr. P.J.Wijkstra, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201700097
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Noninvasive Ventilation
Keywords: COPD; airway inflammation; airway remodeling; health-related auality of life; forced expiratory volume 1 second
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Airway Remodeling | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel groups non-blinded randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NIV directly started arm (Experimental): Patients randomised to this arm will start noninvasive ventilation after baseline measurements are performed.
  Interventions: Device: nocturnal noninvasive ventilation; Other: Standard Care
- NIV postponed arm (Other): Patients randomised to this arm will, after baseline measurements have been done, first be followed for 3 months while on standard care, and thus serve as the control arm. After this 3 months period, measurements are repeated and patients will also be initiated on noninvasive ventilation.
  Interventions: Device: nocturnal noninvasive ventilation; Other: Standard Care

INTERVENTIONS:
Device: nocturnal noninvasive ventilation — Patients will be initiated on bilevel positive pressure non-invasive ventilation via a mask according to regular clinical practice.
Other: Standard Care — Standard COPD care is given to all patients (pharmacological management, oxygen, rehabilitation if neccesary, etc.)

SUMMARY:
Rationale:

Application of long-term non-invasive ventilation (NIV) in chronic obstructive pulmonary disease (COPD) patients with chronic hypercapnic respiratory failure (CHRF) has recently been shown to improve outcomes. However, the mechanism behind these improvements are unknown. We hypothesize that NIV stabilizes FEV1 via beneficial effects on inflammation and repair pathways in patients with COPD. In the present study we aim to investigate, in COPD patients with CHRF,

1. change in FEV1 after 3 months nocturnal NIV in stable hypercapnic COPD patients as compared to standard care
2. the relationship between FEV1 change and modification of systemic and airway inflammation and remodelling, lung hyperinflation, and airway morphology.
3. predictors of a favourable response to chronic NIV in COPD patients with CHRF. Study design: multicentre randomised controlled study investigating the effects of NIV on airway morphology, airway inflammation and remodelling in hypercapnic COPD patients including a control group that will postpone the initiation of NIV for 3 months. In addition we will investigate how patient demographics, patient and disease characteristics and systemic and airway inflammation predict the response to chronic NIV in severe stable COPD. To do this, all patients will be followed for 6 months after NIV initiation.

Main study parameters/endpoints: The main endpoint is the change FEV1 after 3 months. Furthermore, as we recognise that FEV1 might not be the most important patient-related outcome, we will assess which parameters affect health-related quality of life after 3 and 6 months.

DETAILED DESCRIPTION:
Rationale: Application of long-term non-invasive ventilation (NIV) in chronic obstructive pulmonary disease (COPD) patients with chronic hypercapnic respiratory failure (CHRF) has recently been shown to improve outcomes when applied with sufficiently high inspiratory pressures and adequate backup breathing frequencies (high-intensity NIV). Interestingly, it has been demonstrated that nocturnal NIV improves not only clinical but also physiological parameters like arterial carbon dioxide pressure (PaCO¬2¬) and forced expiratory volume in 1 second (FEV1) in patients with stable COPD. However, the mechanism behind these improvements are unknown. Furthermore, it is unclear whether this improvement in lung function influences health-related quality of life (HRQoL), the utmost goal of chronic NIV in COPD, or that other baseline patient- and ventilatory characteristics are more important in predicting a long-term beneficial effect.

We hypothesize that NIV stabilizes FEV1 via beneficial effects on inflammation and repair pathways in the airways of patients with COPD. We aim to study this hypothesis and to investigate the regulation of lung function, markers of inflammation and repair pathways in airway biopsies, bronchial wash and bronchial and nasal epithelium in response to home mechanical ventilation. The second goal of this study is to define a phenotype of patients with COPD, based on baseline characteristics and biomarkers, such as markers of inflammation, who will respond to NIV therapy with improvements in lung function and HRQoL.

Objectives:

1. To investigate change in FEV1 after 3 months nocturnal NIV in stable hypercapnic COPd patients as compared to standard care
2. To investigate the relationship between FEV1 change and modification of systemic and airway inflammation and remodelling, lung hyperinflation, and airway morphology.
3. To investigate predictors of a favourable response to chronic NIV in COPD patients with CHRF.

Study design: The study is multicentre randomised controlled study investigating the effects of NIV on airway morphology, airway inflammation and remodelling in hypercapnic COPD patients including a control group that will postpone the initiation of NIV for 3 months. To measure these parameters a bronchoscopy with a bronchial wash and bronchial biopsies and high-resolution CT-scanning we be done at baseline and after 3 months. In a addition we will investigate how patient demographics, patient and disease characteristics and systemic and airway inflammation predict the response to chronic NIV in severe stable COPD. To do this, all COPD patients initiated on NIV in our centre will be followed for 6 months after NIV initiation as part of the present study.

Study population: Patients who have an indication for NIV (COPD Global Initiative of Obstructive Lung Disease (GOLD) III or IV and a PaCO2 > 6.0 kilopascal (kPa) in stable disease) in the Netherlands will be asked to participate.

For investigating airway inflammation, to ensure safety during the bronchoscopies, patients with severe gas exchange derangements (i.e. PaCO2 > 8.0 kPa and /or partial arterial oxygen pressure (PaO2)<6.5 kPa at rest during spontaneous breathing), and instable cardiac comorbidities will be excluded. These patients will be included to be followed for 6 months prospectively after NIV initiation, according to the same protocol, however, without CT-scanning and bronchoscopies.

Main study parameters/endpoints: The main endpoint is the change FEV1 after 3 months. Several markers of blood and airway inflammation and remodeling will be assessed to analyse mechanisms of FEV1 improvements.

Furthermore, as we recognise that FEV1 might not be the most important patient-related outcome, we will assess which parameters affect health-related quality of life after 3 and 6 months. For this, parameters of the total group of patients will be used.

ELIGIBILITY:
Inclusion Criteria:

* Indication to initiate chronic NIV in COPD patients (GOLD stage III or IV: FEV1/ forced expiratory volume (FVC)< 70% and FEV1< 50% predicted; PaCO2 > 6.0 kilopascal (kPa) in stable condition, which means no COPD exacerbation for 4 weeks and a pH > 7.35)
* Age > 18 years
* Written informed consent is obtained

Exclusion Criteria:

For the randomised Inflammation part a potential subject who meets any of the following criteria will be excluded from participation in this study:

* Oral corticosteroids or roflumilast
* A history of lung volume reduction surgery
* Body mass index (BMI) > 35 kg/m2
* Obstructive sleep apnoea (OSA) (apnoea/hypopnea index (AHI) >15/hr): to exclude OSA a polygraphy will be done at baseline
* PaCO2 ≥ 8.0 kPa or PaO2 < 6.5 kPa at rest without oxygen
* Instable cardiac comorbidities (left ventricular ejection fraction (LVEF) <40%, instable coronary artery disease, instable heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
FEV1 | baseline, 3 months
  Change in Forced expiratory volume in one second
Health-Related Quality of Life | baseline, 3 months, 6 months
  Change in HRQoL assessed by the severe respiratory insufficiency questionnaire summary score (SRI)

SECONDARY OUTCOMES:
Safety: the number of adverse events will be recorded. | baseline, 3 months, and 6 months
  The number of adverse events will be recorded.
Health-related quality of life assessed with the SF-36 | baseline, 3 months, 6 months
  Additional assessment of generic and disease specific aspects of HRQoL, evaluated with the SF-36.
Anxiety and depression | baseline, 3 months, 6 months
  Anxiety and depression, evaluated by the hospital anxiety and depression scale (HADS).
Activities and Restrictions, | baseline, 3 months, 6 months
  Activities and Restrictions, assessed with the Groningen Activity and Restriction Scale (GARS).
Caregiver Burden | baseline, 3 months, 6 months
  Caregiver Burden, assessed with the Caregiver Strain Index (CSI)
Dyspnoea | baseline, 3 months, 6 months
  Dyspnoea, using the Medical Research Council (MRC) score.
Gas exchange day | baseline, 3 months, 6 months
  Gas exchange at daytime without additional oxygen assessed with an arterial blood gas analysis
Gas exchange night | baseline, 3 months, 6 months
  Gas exchange during the night assessed with transcutaneous CO2 measurements.
Respiratory muscle activity | baseline, 3 months
  Respiratory muscle activity during the night and during NIV will be assessed with surface electromyography (EMG)
Spirometry | baseline, 3 months, 6 months
  Spirometry will be used to assess forced expiratory volumes
Exercise tolerance | baseline, 3 months, 6 months
  Exercise tolerance assessed by the 6-minute walking distance.
Peripheral muscle function | baseline, 3 months
  The 1-repetition maximum strength test will performed using a resistance weight-lifting machine
Compliance with the ventilator | baseline, 3 months, 6 months
  Compliance will be read from the ventilator counter readings
Venous blood | Baseline, 3 months
  Venous samples will be obtained for analyses of inflammatory markers
Urine albumin to Creatinine ratio | Baseline, 3 months
  Urine portion for albumin and creatinine will be obtained to obtain the albumin to creatinine ratio
Nasal epithelium markers of remodelling and repair | Baseline, 3 months
  For detailed description see the airway brush markers.
Airway abnormalities | Baseline, 3 months
  Airway abnormalities will be assessed with a High Resolution computertomography (HRCT) scanning with in- and expiration.
Airway inflammation and remodeling | Baseline, 3 months
  Airway inflammation and remodeling assessed with bronchial brushes and washes and airway biopsies obtained through bronchoscopy. Several markers leading to one profile will be assessed
HRQoL assessed with CCQ | Baseline, 3 months, 6 months
  Additional assessment of generic and disease specific aspects of HRQoL, evaluated with the Clinical COPD Questionnaire (CCQ).
Patient-ventilator asynchrony | baseline, 3 months
  Patient-ventilator asynchrony during the night and during NIV will be assessed by comparing surface electromyography (EMG) signals with ventilator pressure tracings
Lung volumes | baseline, 3 months, 6 months
  Bodyplethysmography will be used to assess lung volumes
Emphysema | baseline, 3 months
  The amount of emphysema and air-trapping assessed with a High Resolution computertomography (HRCT) scanning with in- and expiration, and captured into an emphysema score.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Wijkstra, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boersma R, Bakker JT, de Vries M, Raveling T, Slebos DJ, Wijkstra PJ, Hartman JE, Duiverman ML. Defining a phenotype of severe COPD patients who develop chronic hypercapnia. Respir Med. 2024 Nov-Dec;234:107850. doi: 10.1016/j.rmed.2024.107850. Epub 2024 Oct 31. PMID 39488255